CLINICAL TRIAL: NCT05439122
Title: Kinematics and Muscle Performance of the Trunk and Shoulder in Volleyball Players With Subacromial Impingement Syndrome
Status: Completed | Type: Observational
Sponsor: Yi-Fen Shih (Other)
Responsible Party: Sponsor-Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Other Study IDs: YM111061E
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Biomechanical Phenomena
Keywords: Subacromial impingement; muscle performance; volleyball players
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Volleyball players repetitively place the arm into extreme positions, and thus expose the athletes' shoulders to a large load and increase the risk of injuries. The shoulder complex is identified as one of the most injured joints in volleyball sports. Although many studies have revealed alterations in the function, morphology and biomechanics of the shoulder complex in volleyball players with shoulder pain, some researchers suggested that a smooth energy transfer from the axial skeleton, through the shoulder complex, to the arm and hand is crucial for overhead sports performance and injury prevention, with little evidence showing the link between trunk muscle performance and shoulder pain in volleyball players.

Therefore, the main purposes of present study are (1) to compare the trunk muscle performance (muscle strength, power and endurance) in volleyball players with and without subacromial impingement syndrome (SIS); (2) to compare trunk and shoulder muscles activity during spiking in volleyball players with and without SIS.

DETAILED DESCRIPTION:
Volleyball players repetitively place the arm into extreme positions, and thus expose the athletes' shoulders to a large load and increase the risk of injuries. The shoulder complex is identified as one of the most injured joints in volleyball sports. Although many studies have revealed alterations in the function, morphology and biomechanics of the shoulder complex in volleyball players with shoulder pain, some researchers suggested that a smooth energy transfer from the axial skeleton, through the shoulder complex, to the arm and hand is crucial for overhead sports performance and injury prevention, with little evidence showing the link between trunk muscle performance and shoulder pain in volleyball players.

Therefore, the main purposes of present study are (1) to compare the trunk muscle performance (muscle strength, power and endurance) in volleyball players with and without subacromial impingement syndrome (SIS); (2) to compare trunk and shoulder muscles activity during spiking in volleyball players with and without SIS.

We hypothesize that volleyball players with SIS will change in trunk muscle performance and in trunk and shoulder muscles activity during spiking.

This is a cross-sectional case-control exploratory study.The investigators plan to recruit 35 volleyball players with SIS and 35 age, gender, experience matched healthy players in each group, totally 70 volleyball players in this study. Surface electromyography (sEMG) (Noraxon, USA) will be used to collect trunk and shoulder muscles activity during spiking. The kinematics were recorded using the electromagnetic motion tracking system (LIBERTY™). Isokinetic dynamometer (Biodex Multi-Joint System 4 Pro) and (BTE Primus RS) will be used to measure trunk and shoulder muscles torque and power at 60°/s and 180°/s in trunk and 90°/s, 180°/s and 240°/s in shoulder. Flexor, extensor and lateral flexor endurance tests will be used to assess trunk muscles endurance.

SPSS software (version 24.0) will be used to analyze data. The Independent t test or Chi square test will be used to compare demographic data. The Independent two-sample t test will be used to examine group differences in all outcome measures with the significance level setting at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic group:

* The asymptomatic group has to present no history of pain or dysfunction on the shoulder and/or neck in past 6 months.

Subacromial impingement syndrome group:

* Occurrence of shoulder pain that lasted more than 3 months and was related to a spiking movement.
* Present impingement symptoms as a combination of three or more positive signs: Neer test, Hawkins Kennedy test, Jobe test, Painful arc test, Resisted shoulder ER test

Exclusion Criteria:

* Cannot perform spiking movement due to shoulder pain.
* Acute shoulder injury at the time of recruitment or shoulder structural lesion, including hypo/hypermobility, or abnormality.
* History of surgery and fracture in the upper and lower limbs or trunk.
* History of pain in the lower limbs and trunk in the last 3 months.
* Neurological or cardio respiratory disorders.
* Receiving any intervention for the shoulder pain including medication, injection, or general physical therapy during the previous 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Volleyball players with more than 2 years' experience on a collegiate team.
  * Volleyball players have been trained by professional coach over half a year.
  * Playing or training for volleyball over 8 hours per week.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Muscle strength and power of trunk and shoulder | Immediately during the experiment
  The investigator will use isokinetic dynamometer (Biodex Multi-Joint System 4 Pro) and (BTE Primus RS) to measure trunk and shoulder muscles torque and power. Trunk flexion, extension and bilateral rotations will be measured at 60°/s and 180°/s. Shoulder external, internal, horizontal adduction and horizontal abduction will be measured at 90°/s, 180°/s and 240°/s.
Trunk and shoulder muscle activities and kinematics during volleyball spiking | Immediately during the experiment
  The investigator will place surface electromyography (sEMG) (Noraxon, USA) on subjects' bilateral external oblique abdominis, erector spinaes and dominated side of lower trapezius, upper trapezius, serretus anterior and infraspinatus to record muscle activities during spiking. The investigator will also use the electromagnetic motion tracking system (LIBERTY™) to record the kinematics of trunk and shoulder during spiking.
Muscle endurance of trunk and shoulder | Immediately during the experiment
  The subjects will perform trunk flexor, extensor and lateral flexor endurance tests with fixation of lower extremities. The subjects will be asked to hold in a specific position as longer as possible until they quit or fall into wrong position. The holding time will be their score.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided